CLINICAL TRIAL: NCT03399539
Title: Phase I Clinical Trial of Venetoclax (ABT-199) in Combination with Ixazomib and Dexamethasone for Patients with Relapsed Multiple Myeloma
Brief Title: Venetoclax, Ixazomib Citrate, and Dexamethasone in Treating Patients with Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Multiple Myeloma Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC168C; NCI-2017-02456 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC168C (Other: Mayo Clinic); 16-008629 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-01-09; First posted 2018-01-16 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Recurrent Plasma Cell Myeloma; T(11;14)
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ixazomib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (venetoclax, ixazomib citrate, dexamethasone) (Experimental): Patients receive venetoclax PO daily on days 1-28, ixazomib citrate PO once weekly on days 1, 8, and 15, and dexamethasone PO on days 1, 8, 15, and 22 for courses 1-12. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis; Drug: Venetoclax

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta

SUMMARY:
This phase I trial studies the side effects and best dose of venetoclax when given together with ixazomib citrate and dexamethasone and to see how well they work in treating patients with multiple myeloma that has come back. Venetoclax and ixazomib citrate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving venetoclax together with ixazomib citrate and dexamethasone may work better in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of venetoclax in combination with ixazomib citrate (ixazomib) and dexamethasone in patients with relapsed multiple myeloma (MM). (Phase 1)

SECONDARY OBJECTIVES:

I. To describe toxicities associated with venetoclax, in combination with ixazomib and dexamethasone in patients with relapsed MM. (Phase 1)

TERTIARY OBJECTIVES:

I. To explore levels of BCL-2 family member proteins (BCL-2, BCL-x, MCL-1) on bone marrow biopsies using ribonucleic acid sequencing (RNASeq) and immunohistochemistry.

OUTLINE: This is a phase I, dose-escalation study of venetoclax followed by a phase II study.

Patients receive venetoclax orally (PO) daily on days 1-28, ixazomib citrate PO once weekly on days 1, 8, and 15, and dexamethasone PO on days 1, 8, 15, and 22 for courses 1-12. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 or 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1: Relapsed MM with at least one prior line of therapy and should have received a proteasome inhibitor and an immunomodulatory drug
* Phase 2: 1-3 prior lines of therapy and should have received a proteasome inhibitor and an immunomodulatory drug
* Obtained =< 14 days prior to registration: Calculated creatinine clearance (using Cockcroft-Gault equation) >= 30 mL/min
* Obtained =< 14 days prior to registration: Absolute neutrophil count (ANC) >= 1000/uL (without growth factor support)
* Obtained =< 14 days prior to registration: Un-transfused platelet count >= 75000/uL (>= 50,000/uL if marrow plasma cells [PC]% > 50%)
* Obtained =< 14 days prior to registration: Hemoglobin >= 8.0 g/dL
* Obtained =< 14 days prior to registration: Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Obtained =< 14 days prior to registration: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Obtained =< 14 days prior to registration: Alkaline phosphatase =< 750 U/L
* Expansion cohort only: Plasma cell fluorescence in situ hybridization (FISH) test demonstrating presence of t(11;14)
* Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * > 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Provide written informed consent
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willing to follow strict birth control measures as suggested by the study

  * Female patients: If they are of childbearing potential, must agree to one of the following:

    * Practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
  * Male patients: even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

    * Agree to practice effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods and withdrawal are not acceptable methods of contraception)
* Life expectancy >= 12 weeks
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Willing to provide research bone marrow aspirate specimen

Exclusion Criteria:

* Diagnosed or treated for another malignancy =< 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease; NOTE: Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other co-morbidity which would interfere with patient's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease
* Other concurrent chemotherapy or any ancillary therapy considered investigational

  * NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Peripheral neuropathy >= grade 2 on clinical examination or grade 1 with pain during the screening period
* Major surgery =< 14 days prior to study registration
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject?s participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies) or active hepatitis
* Administration of a strong or moderate CYP3A inhibitor or inducer =< 14 days prior to registration
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial
* Failure to have fully recovered (i.e., =< grade 1 toxicity) from the reversible effects of prior chemotherapy
* Radiotherapy =< 14 days prior to registration; Note: If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing
* Previous treatment with ixazomib, or participated in a blinded study with ixazomib
* Live-virus vaccines =< 28 days prior to registration
* Heart failure > New York Heart Association (NYHA) class II

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of venetoclax in combination with ixazomib and dexamethasone (Phase 1) | Up to 28 days
  Defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients (at least 2 of a maximum of 6 new patients). Will be examined in an exploratory and hypothesis-generating fashion.
Overall survival | Time from registration to death due to any cause, assessed up to 3 years
  The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Progression-free survival | Time from registration to the earliest date of documentation of disease progression or death due to any cause, assessed up to 3 years
  The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Rate of confirmed response defined as a patient who has achieved an stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) on two consecutive evaluations (Phase 2) | Up to 3 years
  The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.
Rate of confirmed response in patients with t(11;14) translocation | Up to 3 years
  Will be estimated by the number of patients with a confirmed sCR, CR, VGPR, or PR divided by the total number of evaluable patients with t(11;14) translocation. Exact binomial 95% confidence intervals for the true success proportion will be calculated.
Rate of CR defined as the number of patients with an sCR or CR divided by the total number of evaluable patients | Up to 3 years
  Exact binomial 95% confidence intervals for the true success proportion will be calculated.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 3 years
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Siteman Cancer Center at Washington University, St Louis, Missouri

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials